CLINICAL TRIAL: NCT05107921
Title: Efficacy of Bromfenac Sodium Hydrate Eye Drops in Children With Familial Exudative Vitreoretinopathy After Diode Laser Photocoagulation
Brief Title: Bromfenac Sodium Hydrate Eye Drops in Familial Exudative Vitreoretinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Hun Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2107-210-1239
Record Dates: First submitted 2021-10-23; First posted 2021-11-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Familial Exudative Vitreoretinopathies
MeSH Terms: conditions — Familial Exudative Vitreoretinopathies | interventions — bromfenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bromfenac sodium hydrate eye drops (Experimental): The patients will receive bromfenac sodium hydrate eye drops twice daily for 14 days.
  Interventions: Drug: Bromfenac Sodium

INTERVENTIONS:
Drug: Bromfenac Sodium — The study participants will receive bromfenac sodium hydrate eyedrops twice daily for 14 days.
  Other Names: Bronuck

SUMMARY:
This study aims to investigate the efficacy and safety of bromfenac sodium hydrate eye drops in patients with familial exudative vitreoretinopathy receiving diode laser photocoagulation.

DETAILED DESCRIPTION:
This study aims to evaluate the presence of macular edema as the primary measure and the presence of conjunctival injection as the secondary measure for the investigation of the efficacy of bromfenac sodium hydrate eye drops in patients with familial exudative vitreoretinopathy receiving diode laser photocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with familial exudative vitreoretinopathy
* Needing diode laser photocoagulation
* Consent to the study

Exclusion Criteria:

* History of corneal diseases
* History of hypersensitivity to bromfenac sodium
* History of hypersensitivity to non-steroidal anti-inflammatory drugs
* Progressive ocular infection
* Liver diseases
* Hypersensitivity to sulfur dioxide
* Receiving anti-coagulation drugs
* History of coagulopathies

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Macular edema response rate | 4 weeks after the diode laser photocoagulation
  Presence of macular edema

SECONDARY OUTCOMES:
Conjunctival injection response rate | 4 weeks after the diode laser photocoagulation
  Presence of conjunctival injection

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hun Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No